CLINICAL TRIAL: NCT02990104
Title: Diagnostic and Treatment in Acute Lymphoblastic Leukemia Adults: A Multicenter Study of Five Years Experience, Retrospective in Acute Lymphoblastic Leukemia Adults Patients, Mexico City: First Report of the Acute Leukemia Work Group (GTLA)
Brief Title: First Report, Five Years Experience of the Acute Leukemia Work Group
Acronym: PR-GTLA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mexican Agrupation for Hematology Study (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 2016001/PR-GTLA
Record Dates: First submitted 2016-12-05; First posted 2016-12-13 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-11

CONDITIONS: Acute Leukemia (Category)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to describe the incidence, clinic characteristics, biological and suvirval in Lymphoblastic Leukemia patients in Mexico City reference hospitals.

DETAILED DESCRIPTION:
Multicenter and retrospective revision of clinical files with Acute Lymphoblastic Leukemia diagnostic between 2009 and 2013 in Mexico City reference hospitals, in five hospitals with 50 and 100 new cases Acute Lymphoblastic Leukemia per year. With a expected sample between 500 and 1000 patients it will descriptive statistics of variables. The data collection with necessary variables for survival analysis study and risk factors with Kaplan-Meier curve and risk proportional method Cox.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Acute Lymphoblastic Leukemia

Exclusion Criteria none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute Lymphoblastic Leukemia
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-01 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Get the incidence of Acute Lymphoblastic Leukemia in Mexico City reference hospitals | 5 years
  Date collection from clinical files with Acute Lymphoblastic Leukemia diagnostic between 2009 and 2013 in Mexico City in 5 reference hospitals

SECONDARY OUTCOMES:
Clinic characteristics, biological and survival in Acute Lymphoblastic Leukemia patients in Mexico City reference hospitals | 5 years
  Date collection from clinical files with Acute Lymphoblastic Leukemia diagnostic between 2009 and 2013 in Mexico City in 5 reference hospitals

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Erick Crespo, Doctor, Principal Investigator — Regional Hospital High Speciality, Tamaulipas Cd. Victoria
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico Distrito Federal, Mexico

IPD SHARING:
Plan to Share IPD: Undecided